CLINICAL TRIAL: NCT03724812
Title: Assessment of the Abbott FlexNav™ Delivery System for Portico Transcatheter Aortic Valve Implantation in High and Extreme Risk Patients With Symptomatic Severe Aortic Stenosis
Brief Title: FlexNav EU CE Mark Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10260
Record Dates: First submitted 2018-10-29; First posted 2018-10-30 (Actual); Results first posted 2021-03-16 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-10

CONDITIONS: Symptomatic Severe Aortic Stenosis
Keywords: Aortic Stenosis; FlexNav™ Delivery System; Portico Delivery System; Transcatheter Aortic Valve Replacement; Heart Valve Disease; High surgical risk
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases

STUDY DESIGN:
Intervention Model Description: Devices under investigation in this clinical investigation include the FlexNav™ Delivery System(s) (18 F and 19 F) and FlexNav™ Loading System(s) (Small and Large), which are both approved for investigational use only. Other devices to be used in the clinical investigation include all four (4) market released Abbott Portico™ valve sizes (23mm, 25mm, 27mm and 29mm).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Portico valve and FlexNav™ Delivery System (Experimental): Portico valve implantation with the second-generation FlexNav Delivery system
  Interventions: Device: Portico Valve and FlexNav™ Delivery System

INTERVENTIONS:
Device: Portico Valve and FlexNav™ Delivery System — Subjects will undergo transcatheter aortic valve replacement (TAVR) with the Portico valve and second-generation FlexNav Delivery system via a transfemoral access approach

SUMMARY:
The purpose of this clinical investigation is to characterize the safety of the next-generation FlexNav™ Delivery System for transfemoral implantation of the Portico™ Transcatheter Aortic Heart Valve in symptomatic severe aortic stenosis patients who are considered of high or extreme risk for surgical aortic valve replacement. Data from the study will be used to support CE Mark of the FlexNav™ Delivery System and Loading System in Europe.

DETAILED DESCRIPTION:
The FlexNav European Union (EU) study will be conducted as a prospective, multi-center, single-arm investigational study.

High or extreme risk patients with symptomatic, severe native aortic stenosis who are determined by an independent subject selection committee to meet eligibility criteria for Portico™ Transcatheter Aortic Heart Valve implantation via a transfemoral access approach will undergo a Portico valve implant using the next-generation FlexNav Delivery System.

Subject data will be collected at screening, baseline, pre-procedure, peri-procedure, post-procedure, discharge, 30 days, 6 months and 1-year from the index procedure.

ELIGIBILITY:
Inclusion Criteria:

- Candidates for High Risk classification must meet all the following inclusion criteria:

1. Subjects must have co-morbidities such that the local heart team concur the predicted risk of operative mortality is ≥15% or a minimum Society of Thoracic Surgeons (STS) score of 8%.

   a) A candidate who does not meet the STS score criteria of ≥ 8% may be included in the study if at least one surgeon in the local heart team concludes and documents the patient's predicted risk of operative mortality is ≥15%. The surgeon's assessment of operative comorbidities (including frailty indices) not captured by the STS score must be documented in the study case report form as well as in the patient medical record.
2. Subject is of legal age or older for consent in the host country.
3. Subject has senile degenerative aortic valve stenosis with echo-derived criteria: mean gradient >40 mmHg or jet velocity greater than 4.0 m/s or doppler velocity index (DVI) <0.25 and an initial aortic valve area (AVA) of ≤1.0 cm2 (indexed Effective Orifice Area (EOA) ≤ 0.6 cm2/m2). (Qualifying AVA baseline measurement must be within 60 days prior to informed consent).
4. Subject has symptomatic aortic stenosis as demonstrated by NYHA Functional Classification of II, III, or IV.
5. The subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board (IRB) of the respective clinical site.
6. The subject and the treating physician agree that the subject will return for all required post-procedure follow-up visits.
7. Subject's aortic annulus is 19-27mm diameter as measured by computed tomography (CT) conducted within 12 months prior to informed consent. If a CT i contraindicated and/or not possible to be obtained for certain subjects, a 3D echo and non-contrast CT of chest and abdomen/pelvis may be accepted.

   All candidates for Extreme Risk classification must meet # 2, 3, 4, 5, 6, 7 of the above criteria, and
8. After formal consultation with the local heart team (including at least one surgeon) it is agreed that medical factors preclude the subject from undergoing operation, based on a conclusion that the probability of death or serious, irreversible morbidity exceeds the probability of meaningful improvement. Specifically, the probability of death or serious, irreversible morbidity should exceed 50%. The local heart teams' consult notes shall specify the medical or anatomic factors leading to that conclusion and include a printout of the calculation of the STS score to additionally identify the risks in these patients.

Exclusion Criteria:

Candidates will be excluded if any of the following conditions are present:

1. Evidence of an acute myocardial infarction (defined as: ST Segment Elevation as evidenced on 12 Lead ECG) within 30 days prior to index procedure.
2. Aortic valve is a congenital unicuspid or congenital bicuspid valve, or is noncalcified as verified by echocardiography.
3. Mixed aortic valve disease (aortic stenosis and aortic regurgitation with predominant aortic regurgitation 3-4+).
4. Any percutaneous coronary or peripheral interventional procedure performed within 30 days prior to index procedure.
5. Pre-existing prosthetic heart valve or other implant in any valve position, prosthetic ring, severe circumferential mitral annular calcification (MAC) which is continuous with calcium in the LVOT, severe (greater than 3+) mitral insufficiency, or severe mitral stenosis with pulmonary compromise.
6. Blood dyscrasias as defined: leukopenia (WBC<3000 mm3), acute anemia (Hb < 9 g/dL), thrombocytopenia (platelet count <50,000 cells/mm³).
7. History of bleeding diathesis or coagulopathy.
8. Cardiogenic shock manifested by low cardiac output, vasopressor dependence, or mechanical hemodynamic support.
9. Untreated clinically significant coronary artery disease requiring revascularization.
10. Hemodynamic instability requiring inotropic support or mechanical heart assistance.
11. Need for emergency surgery for any reason.
12. Hypertrophic cardiomyopathy with or without obstruction (HOCM).
13. Severe ventricular dysfunction with left ventricular ejection fraction (LVEF) <20% as measured by resting echocardiogram.
14. Echocardiographic evidence of intracardiac mass, thrombus or vegetation.
15. Active peptic ulcer or upper GI bleeding within 3 months prior to index procedure.
16. A known hypersensitivity or contraindication to aspirin, heparin, ticlopidine (Ticlid), or clopidogrel (Plavix), or sensitivity to contrast media which cannot be adequately premedicated.
17. Recent (within 6 months prior to index procedure date) cerebrovascular accident (CVA) or a transient ischemic attack (TIA).
18. Renal insufficiency (creatinine > 3.0 mg/dL) and/or end stage renal disease requiring chronic dialysis.
19. Life expectancy < 12 months from the time of informed consent due to noncardiac co-morbid conditions.
20. Significant aortic disease, including abdominal aortic or thoracic aneurysm defined as maximal luminal diameter 5cm or greater; marked tortuosity (hyperacute bend), aortic arch atheroma (especially if thick [> 5 mm], protruding or ulcerated) or narrowing (especially with calcification and surface irregularities) of the abdominal or thoracic aorta, severe "unfolding" and tortuosity of the thoracic aorta.
21. Native aortic annulus size < 19 mm or > 27 mm per the baseline diagnostic imaging.
22. Aortic root angulation > 70°.
23. Currently participating in an investigational drug or device study.
24. Active bacterial endocarditis within 6 months prior to the index procedure.
25. Bulky calcified aortic valve leaflets in close proximity to coronary ostia.
26. Non-calcified aortic annulus.
27. Iliofemoral vessel characteristics that would preclude safe insertion of the FlexNav™ delivery system with or without an arterial introducer sheath such as severe obstructive calcification, or severe tortuosity.
28. In the judgment of the investigator, a condition that could limit a patient's ability or willingness to participate in the study, comply with study required testing and/or follow- up visits or that could impact scientific integrity of the study.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2021-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Bedogni, MD, Principal Investigator — Policlinico San Donato
Locations (6):
- Rigshospitalet, Copenhagen, Denmark
- Policlinico San Donato, San Donato Milanese, Lombard, Italy
- Switzerland (2):
  - Kantonsspital St. Gallen, Sankt Gallen
  - Universitaets Spital Zuerich, Zurich
- United Kingdom (2):
  - Morriston Hospital - ABM University Health Board, Morriston, Swansea
  - Royal Victoria Hospital, Belfast

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between 26 February 2019 and 10 December 2019
Groups:
- Portico Valve and FlexNav™ Delivery System: Subjects will undergo an attempted transcatheter aortic valve replacement (TAVR) with the Portico valve and next-generation FlexNav Delivery system via a transfemoral access approach
Period: Overall Study
Arm/Group | Portico Valve and FlexNav™ Delivery System
Started | 46
Discharge | 46
30 Day Follow-Up | 45
6 Month Follow-Up | 42
12-Month Follow-Up | 42
Completed | 42
Not Completed | 4
Not completed — Missed Visit | 1
Not completed — Death | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Analysis population includes subjects that underwent an attempted Portico valve implant with the FlexNav delivery system
Arm/Group | Portico Valve and FlexNav™ Delivery System
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 85.4 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Denmark | 3
  Italy | 17
  United Kingdom | 22
  Switzerland | 4

OUTCOME MEASURES:

1. Primary Outcome: Major Vascular Complications
Description: Percentage of patients with a VARC-2 defined major vascular complication event
Time Frame: At 30 days post index procedure
Population: Analysis population included all subjects in whom a Portico valve implant was attempted (enrolled subjects)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Portico Valve and FlexNav™ Delivery System: Subjects that underwent an attempted transcatheter aortic valve replacement (TAVR) with the Portico valve and FlexNav Delivery system via a transfemoral access approach
Arm/Group | Portico Valve and FlexNav™ Delivery System
Number analyzed (Participants) | 46
percentage of participants | 4.3 [0.5 to 14.8]

2. Other Pre Specified Outcome: Non-hierarchical Composite Safety Endpoint
Description: Percentage of patients with a non-hierarchical composite endpoint of all-cause mortality, disabling stroke, life threatening bleeding requiring blood transfusion, acute kidney injury requiring dialysis, or major vascular complications
Time Frame: 30 days from the index procedure.
Population: Analysis population included all subjects in whom a Portico valve implant was attempted (enrolled subjects)
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Portico Valve and FlexNav™ Delivery System
Number analyzed (Participants) | 46
percentage of subjects | 6.5 [1.37 to 17.90]

3. Other Pre Specified Outcome: All-Cause Mortality
Description: Percentage of patients with VARC 2 defined all-cause mortality
Time Frame: 30 days from the index procedure
Population: Analysis population included all subjects in whom a Portico valve implant was attempted (enrolled subjects)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Portico Valve and FlexNav™ Delivery System
Number analyzed (Participants) | 46
percentage of participants | 0 [0.0 to 7.71]

4. Other Pre Specified Outcome: Disabling Stroke
Description: Percentage of patients with a VARC-2 defined disabling stroke event
Time Frame: 30 days from index procedure
Population: Analysis population included all subjects in whom a Portico valve implant was attempted (enrolled subjects)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Portico Valve and FlexNav™ Delivery System
Number analyzed (Participants) | 46
percentage of participants | 0 [0.0 to 7.71]

5. Other Pre Specified Outcome: Life-threatening Bleeding Requiring Blood Transfusion
Description: Percentage of patients with a VARC-2 defined life-threatening bleeding event requiring blood transfusion
Time Frame: 30 days from the index procedure
Population: Analysis population included all subjects in whom a Portico valve implant was attempted (enrolled subjects)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Portico Valve and FlexNav™ Delivery System
Number analyzed (Participants) | 46
percentage of participants | 4.3 [0.53 to 14.84]

6. Other Pre Specified Outcome: Major Bleeding Event
Description: Percentage of patients with VARC 2 defined major bleeding event
Time Frame: 30 days from index procedure
Population: Analysis population included all subjects in whom a Portico valve implant was attempted (enrolled subjects)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Portico Valve and FlexNav™ Delivery System
Number analyzed (Participants) | 46
percentage of participants | 4.3 [0.53 to 14.84]

7. Other Pre Specified Outcome: Acute Kidney Injury
Description: Percentage of patients with a VARC 2 defined acute kidney injury event
Time Frame: 30 days from index procedure
Population: Analysis population included all subjects in whom a Portico valve implant was attempted (enrolled subjects)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Portico Valve and FlexNav™ Delivery System
Number analyzed (Participants) | 46
percentage of participants | 0 [0.0 to 7.71]

8. Other Pre Specified Outcome: Minor Vascular Complication
Description: Percentage of patients with a VARC-2 defined minor vascular complication
Time Frame: 30 days from index procedure
Population: Analysis population included all subjects in whom a Portico valve implant was attempted (enrolled subjects)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Portico Valve and FlexNav™ Delivery System
Number analyzed (Participants) | 46
percentage of participants | 15.2 [6.34 to 28.87]

9. Other Pre Specified Outcome: New Permanent Pacemaker Implant
Description: Percentage of patients requiring a new permanent pacemaker. Excludes patients with a pre-existing permanent pacemaker at baseline
Time Frame: 30 days from index procedure
Population: Analysis population included all subjects in whom a Portico valve implant was attempted (enrolled subjects) and who did not have a pre-existing pacemaker at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Portico Valve and FlexNav™ Delivery System: Subjects without a permanent pacemaker at baseline that underwent an attempted transcatheter aortic valve replacement (TAVR) with the Portico valve and FlexNav Delivery system via a transfemoral access approach
Arm/Group | Portico Valve and FlexNav™ Delivery System
Number analyzed (Participants) | 42
percentage of participants | 14.3 [5.43 to 28.54]

10. Other Pre Specified Outcome: Severity of Paravalvular Leak
Description: Echocardiographic core-laboratory derived severity of paravalvular leak
Time Frame: 30 days from index procedure
Population: Analysis population included all subjects in whom a Portico valve implant was attempted (enrolled subjects) with an analyzable echocardiogram at 30 days
Measure: Number; unit: percentage of patients
Arm/Group | Portico Valve and FlexNav™ Delivery System
Number analyzed (Participants) | 43
percentage of patients
  None/Trace/Trivial PVL | 53.5
  Mild PVL | 46.5
  Moderate PVL | 0
  Severe PVL | 0

11. Other Pre Specified Outcome: NYHA Functional Classification
Description: Proportion of subjects with a NYHA Functional Class of I,II, III or IV (range I-IV where a lower score indicates less limitation in physical activity)
Time Frame: 30 days from index procedure
Population: Analysis population included all subjects in whom a Portico valve implant was attempted (enrolled subjects). Information was not available for one subject.
Measure: Number; unit: percentage of participants
Arm/Group | Portico Valve and FlexNav™ Delivery System
Number analyzed (Participants) | 45
percentage of participants
  NYHA I | 48.9
  NYHA II | 48.9
  NYHA III | 2.2
  NYHA IV | 0

12. Other Pre Specified Outcome: Kansas City Cardiomyopathy Questionnaire Quality of Life (QOL) Score
Description: KCCQ Overall summary score (range 0-100 where a higher score indicates a better quality of life and physical function)
Time Frame: 30 days from index procedure
Population: Analysis population included all subjects in whom a Portico valve implant was attempted (enrolled subjects). Information was not available for 2 subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Portico Valve and FlexNav™ Delivery System
Number analyzed (Participants) | 44
score on a scale | 66.46 (20.86)

13. Other Pre Specified Outcome: Technical Device Success
Description: Technical device success defined as successful vascular access, delivery and deployment of the Portico Valve; retrieval with the delivery system and correct positioning of a single valve in the proper anatomical location.
Time Frame: Over the duration of index procedure, an average of 60.6 minutes
Population: Analysis population included all subjects in whom a Portico valve implant was attempted (enrolled subjects)
Measure: Number; unit: percentage of participants
Arm/Group | Portico Valve and FlexNav™ Delivery System
Number analyzed (Participants) | 46
percentage of participants | 100

14. Other Pre Specified Outcome: All-Cause Mortality or Disabling Stroke
Description: Percentage of patients with a composite of all-cause mortality or disabling stroke at one year from the index procedure censored for COVID-19 related events
Time Frame: One year (365 days) from index procedure
Population: sensitivity analyses censoring subject's first COVID-19 related endpoint event
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Portico Valve and FlexNav™ Delivery System
Number analyzed (Participants) | 46
percentage of participants | 2.2 [0.32 to 14.75]

15. Other Pre Specified Outcome: All-Cause Mortality
Description: Percentage of patients that died at one year from the index procedure censored for COVID-19 related endpoint events
Time Frame: One year (365 days) from index procedure
Population: sensitivity analyses censoring subject's first COVID-19 related endpoint event
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Portico Valve and FlexNav™ Delivery System
Number analyzed (Participants) | 46
percentage of participants | 2.2 [0.32 to 14.75]

16. Other Pre Specified Outcome: Disabling Stroke
Description: Percentage of patients with a disabling stroke at one year from index procedure censored for COVID-19 related endpoint events
Time Frame: One Year (365 days) from index procedure
Population: sensitivity analyses censoring subject's first COVID-19 related endpoint event
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Portico Valve and FlexNav™ Delivery System
Number analyzed (Participants) | 46
percentage of participants | 0 [0 to 0]

17. Other Pre Specified Outcome: Severity of Paravalvular Leak
Description: Echocardiographic core-laboratory derived severity of paravalvular leak
Time Frame: One year from index procedure
Population: as for outcome 10
Measure: Number; unit: percentage of patients
Arm/Group | Portico Valve and FlexNav™ Delivery System
Number analyzed (Participants) | 36
percentage of patients
  None/Trace/Trivial PVL | 72.2
  Mild PVL | 27.8
  Moderate PVL | 0.0
  Severe PVL | 0.0

18. Other Pre Specified Outcome: NYHA Functional Classification
Description: as for outcome 11
Time Frame: One year from index procedure
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Portico Valve and FlexNav™ Delivery System
Number analyzed (Participants) | 40
percentage of participants
  NYHA I | 57.5
  NYHA II | 40.0
  NYHA III | 2.5
  NYHA IV | 0.0

19. Other Pre Specified Outcome: Kansas City Cardiomyopathy Questionnaire Quality of Life (QOL) Score
Description: KCCQ Overall summary score (range 0-100 where a higher score indicates a better quality of life and physical function)
Time Frame: One year from index procedure
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Portico Valve and FlexNav™ Delivery System
Number analyzed (Participants) | 40
score on a scale | 71.11 (16.71)

ADVERSE EVENTS:
Time Frame: Site-reported adverse events related to the investigational study device within 1 year follow-up
Arm/Group | Portico Valve and FlexNav™ Delivery System
All-Cause Mortality (participants affected / at risk) | 2/46
Serious Adverse Events (participants affected / at risk) | 21/46
Other Adverse Events (participants affected / at risk) | 19/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Portico Valve and FlexNav™ Delivery System (N=46)
Arrhythmias (Cardiac disorders) | 3 (4)
Endocarditis (Cardiac disorders) | 1 (2)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1)
Pericardial Tamponade (Cardiac disorders) | 1 (1)
Heart Block (Cardiac disorders) | 5 (5)
Heart Failure (Cardiac disorders) | 5 (6)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Bacterial Infection (Infections and infestations) | 2 (3)
General (General disorders) | 10 (12)
Stroke (Nervous system disorders) | 2 (2)
Vascular Access Site Complications (Injury, poisoning and procedural complications) | 2 (2)
Coronary Artery Disease (Cardiac disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
Bleeding (General disorders) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 2 (2)
General-Musculoskeletal Symptoms (Musculoskeletal and connective tissue disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (3)
Seizure/Convulsions/Epilepsy (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Portico Valve and FlexNav™ Delivery System (N=46)
Arrhythmias (Cardiac disorders) | 4 (4)
Arterial Hypertension (Cardiac disorders) | 1 (1)
Heart Block (Cardiac disorders) | 10 (10)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Anemias (Blood and lymphatic system disorders) | 5 (5)
Bleeding (Blood and lymphatic system disorders) | 1 (1) — General
Hematoma (Blood and lymphatic system disorders) | 2 (2) — General
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Allergy (General disorders) | 1 (1)
Other (General disorders) | 7 (10)
Dental Disorders (General disorders) | 1 (1)
Thyroid Disorders (Endocrine disorders) | 1 (1)
Edema (Renal and urinary disorders) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
Aortic Valve Regurgitation/Aortic Valve Insufficiency/Valvular Regurgitation Aortic Valve (Product Issues) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-10-23): https://cdn.clinicaltrials.gov/large-docs/12/NCT03724812/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT03724812/SAP_001.pdf